CLINICAL TRIAL: NCT04174209
Title: CHOICE OF SUBJECTIVE OCULAR REFRACTION TECHNIQUE AND CORNEAL TOPOGRAPHY OF KERATOCONUS
Acronym: RE-CON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 CHIAMBARETTA; 2019-A01624-53 (Other: 2019-A01624-53)
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2019-11

CONDITIONS: Keratoconus; Alteration of Visual Acuity
Keywords: Keratoconus; Corneal Topography; Eyeglasses; Ocular Refraction; Jackson Cross Cylinder; Astigmatic Dial Technique; Stenopeic slit
MeSH Terms: conditions — Keratoconus | interventions — cylindrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): 70 patients are involved and will perform the three conditions.
  Interventions: Behavioral: Cylinder; Behavioral: Dial; Behavioral: Slit

INTERVENTIONS:
Behavioral: Cylinder — Patients who receive the Jackson Cross Cylinder Method
Behavioral: Dial — Patients who receive the Astigmatic Dial Technique Method.
Behavioral: Slit — Patients who receive the Stenopeic slit Method.

SUMMARY:
Keratoconus is a rare evolving corneal ectasia that alters visual acuity. To improve spectacle-corrected visual acuity, various subjective refraction techniques can be used.

The subjective refraction techniques of keratoconus-carrying patients have never been studied.

The main hypothesis is that the most suitable subjective ocular refraction method varies with the corneal topography of the keratoconus.

The main objective is to define the most appropriate refractive technique(s) based on corneal topographies in order to provide keratoconus-affected patients with the best spectacle-corrected visual acuity.

DETAILED DESCRIPTION:
Keratoconus is a rare evolving corneal ectasia that alters visual acuity. To improve spectacle-corrected visual acuity, various subjective refraction techniques can be used. The Jackson Cylinder Cross Method, the Astigmatic Dial Technique and the Stenopeic Slit are three validated subjective refraction techniques for measuring astigmatism. The subjective refraction techniques of keratoconus-carrying patients have never been studied.

The main hypothesis is that the most suitable subjective ocular refraction method varies with the corneal topography of the keratoconus.

The investigators collect several characteristics of corneal topography of the keratoconus : the average value of the keratometry of the 3 central mm called Km ; the value of the point corresponding to the maximum keratometry (called Kmax), the distance between the center and the point of Kmax, (called d_Kmax) ; the corneal surface variance index called ISV ; the Belin/Ambrósio Enhanced Ectasia Display (called BAD-D).

The main objective is to define the most appropriate refractive technique(s) based on corneal topographies in order to provide keratoconus-affected patients with the best spectacle-corrected visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* adult persons
* patients with keratoconus
* patients with alteration of visual acuity
* ability to give informed consent to participate in the study
* affiliation to a social security scheme

Exclusion Criteria:

* Keratoconus grafted with cornea or with intracorneal rings.
* Central corneal opacities.
* Presence of other eye diseases affecting visual acuity.
* Patients under guardianship, curatorship or justice protection.
* Pregnant or breastfeeding women.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Measure of keratometry (Km) | day 1
  average value of the keratometry of the 3 central mm called Km
Measure of the maximum keratometry | day 1
  value of the point corresponding to the maximum keratometry (called Kmax),
Measure d_Kmax | day 1
  Measure of the distance between the center and the point of Kmax, (called d_Kmax)
Measure of index of surface varaiance | day 1
  measure of the corneal surface variance index called ISV
Measure of the Belin/Ambrósio Enhanced Ectasia Display (BAD-D) | day 1
  Measure of the Belin/Ambrósio Enhanced Ectasia Display (BAD-D)

SECONDARY OUTCOMES:
astigmatism axis | day 1
  Collection of the astigmatism axis given by each method, by the autorefractometer and by the corneal topography
Subsequent modification of the eyeglasses by the optician | day 30
  The need (yes / no) for the optician to modify the prescribed spectacle lens (due to poor tolerance)
possible method | day 1
  The impossibility (yes / no) of carrying out each of the 3 refraction methods.
ametropia value | day 1
  The values of the final corrective spheres (myopia or hyperopia).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Chiambaretta, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Metzger M, Navel V, Barriere JV, Kwiatkowski F, Hebraud J, Mulliez A, Beral L, Chiambaretta F, Dutheil F. Benefits of using corneal topography to choose subjective refraction technique in keratoconus (RE-CON): a prospective comparative crossover clinical study. Graefes Arch Clin Exp Ophthalmol. 2022 Jan;260(1):197-207. doi: 10.1007/s00417-021-05382-y. Epub 2021 Aug 20. PMID 34415365